CLINICAL TRIAL: NCT02185651
Title: A Pilot Study of the Effects of Oral Administration of Zavesca® on Anti-rhGAA Immune Response in Subjects With Pompe Disease Receiving rhGAA Enzyme Replacement Therapy
Brief Title: A Pilot Study of Zavesca® in Patients With Pompe Disease and Infusion Associated Reaction
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Participants not interested in enrolling.
Sponsor: University of Florida (Other)
Collaborators: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601641
Record Dates: First submitted 2014-07-01; First posted 2014-07-09 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Pompe Disease; Hypersensitivity Reaction
Keywords: Pompe Disease; Enzyme Replacement Therapy; Infusion Associated Reaction
MeSH Terms: conditions — Glycogen Storage Disease Type II; Hypersensitivity | interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zavesca® 100 mg (Active Comparator): 3 study participants are given Zavesca® prescription 100 mg for administration before ERT infusion. Week 0 infusion is completed at study site, with blood collection for anti-GAA antibody level before, during and after the ERT infusion. A punch muscle biopsy is completed the day after ERT infusion with pre-medication Zavesca®. Health Survey is completed.
  Week 2, 4, and 6 ERT infusion with pre-medication are completed at local/home infusion center. Travel to site for week 7 study visit includes physical exam, blood collection and punch muscle biopsy. Health survey is completed.
  Interventions: Drug: Zavesca® Prescription
- Zavesca® 300 mg (Active Comparator): 3 study participants are given Zavesca® prescription 300 mg for administration before ERT infusion. Week 0 infusion is completed at study site, with blood collection for anti-GAA antibody level before, during and after the ERT infusion. A punch muscle biopsy is completed the day after ERT infusion with pre-medication Zavesca®. Health Survey is completed.
  Week 2, 4, and 6 ERT infusion with pre-medication are completed at local/home infusion center. Travel to site for week 7 study visit includes physical exam, blood collection and punch muscle biopsy. Health survey is completed.
  Interventions: Drug: Zavesca® Prescription

INTERVENTIONS:
Drug: Zavesca® Prescription — Following baseline evaluation, Zavesca® prescription is given.
  Week 2, 4, and 6 ERT infusion with pre-medication are completed at local/home infusion center. Travel to site for week 7 study visit includes physical exam, blood collection and punch muscle biopsy. Health survey is completed.
  Other Names: miglustat

SUMMARY:
Hypothesis: the effectiveness of treatment of Pompe disease with rhGAA enzyme replacement therapy (ERT) is limited at least in part because patients develop antibodies against the provided rhGAA enzyme. Treatment with Zavesca® prior to infusion may dampen or eliminate the anti-rhGAA immune response in patients receiving ERT, thereby allowing for greater ERT efficacy.

Treatment with Zavesca® before a enzyme replacement therapy (ERT) may decrease the severity of, or eliminate infusion associated reactions (IAR) in people with Pompe Disease receiving ERT.

DETAILED DESCRIPTION:
This Study is designed to assess the effects of Zavesca® as immunomodulatory therapy on anti-rhGAA immune responses in patients with Pompe disease, as well as their health and disease progression. Subjects will either receive Zavesca® at 100 mg or 300 mg dosing levels during study participation (n=3 @ 100 mg dosing; n=3 @ 300 mg dosing).

The first 3 subjects enrolled will be prescribed 100 mg Zavesca® 60 minutes prior to ERT infusion. The subsequent 3 subjects enrolled will be prescribed 300 mg Zavesca® 60 minutes to ERT infusion.

Eligible participants are on standard ERT for Pompe disease and have a history of infusion associated reaction. Travel to the study site in Gainesville, Florida is required for 3 visits. Participants are prescribed medication Zavesca® and have blood tests, punch muscle biopsy, physical exams, and answer questionnaires over 3 months study participation.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be patients between the ages of 18 years and 65 years who have been diagnosed with Pompe Disease, confirmed by mutational analysis and/or GAA enzyme activity assay.

* Receiving rhGAA ERT
* Willing to travel to the study site for study assessments
* Willingness of local medical treatment provider to continue treating study participant with addition of Zavesca® to treatment plan.
* Willingness of study participant to modify dietary intake on day of infusion *All Subjects will continue enzyme replacement therapy as standard of care, as prescribed by local medical treatment provider during the course of the Study.

Exclusion Criteria:

* Subject is unable to meet the study requirements
* Subject's medical condition contraindicates participation or Study Investigators feel that participation is otherwise not in the Subject's best interest
* Subject does not receive ERT treatment
* Participation in other interventional studies at the time of enrollment that may interfere with this study (at the investigator's discretion)
* Unable to travel to the University of Florida for study visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Evaluate Pharmacodynamics of ERT with pre-medication Zavesca | Baseline, week 0, week 6
  Change in GAA antibody level from Baseline to week 0: GAA antibody titer is reported at timepoints: pre-infusion, and 6, 12, and 24 hours post-infusion start.
  Change in GAA antibody level from Baseline to week 6: GAA antibody titer is reported at time points: pre-infusion and post-infusion.

SECONDARY OUTCOMES:
Evaluate pharmacokinetics of ERT with pre-medication Zavesca® | Baseline, week 0
  Change in ERT half life at baseline (without Zavesca®) compared to week 0 (ERT with pre-medication Zavesca®).
  Change in Maximum plasma concentration (Cmax) at baseline (without Zavesca®) compared to week 0 (ERT with pre-medication Zavesca®).
Evaluate biodistribution of ERT with pre-medication Zavesca®. | Week 0, week 7
  Punch muscle biopsy is performed at week 0 and week 7 for biodistribution: Change in glycogen content and muscle fiber morphology is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Barry J. Byrne, MD, PhD, Principal Investigator — University of Florida